CLINICAL TRIAL: NCT06655103
Title: The Effect of the Educational Movie Shown to Pediatric Patients Receiving Intrathecal Chemotherapy Treatment on Pre-Procedure Fear and Post-Procedure Pain in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Aycin Ezgi ONEL, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EGEUNIVERSITY-ONEL-001
Record Dates: First submitted 2024-10-19; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Injections, Spinal; Child, Only; Virtual Reality; Fear; Pain; Chemotherapy
Keywords: Intrathecal; Child; Virtual reality; Fear; Pain; chemotherapy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group shown educational movie with virtual reality glasses (Experimental): Measurements will be performed in three stages. In the first measurement; electrodermal activity, pulse, respiration and oxygen (O2) saturation values together with fear and pain scales 30 minutes before IT chemotherapy treatment without any intervention, in the second measurement; Electrodermal activity, pulse, respiration and O2 saturation values together with fear and pain scales after the application of virtual reality goggles 15 minutes before IT chemotherapy, and in the third measurement, electrodermal activity, pulse, respiration and O2 saturation values together with fear and pain scales will be evaluated within 30-60 minutes after IT chemotherapy treatment (when the sedation effect is over).
  Interventions: Other: Educational movie
- Group watching cartoons with virtual reality glasses (Experimental): Measurements will be performed in three stages. In the first measurement; electrodermal activity, pulse, respiration and oxygen (O2) saturation values together with fear and pain scales 30 minutes before IT chemotherapy treatment without any intervention, in the second measurement; Electrodermal activity, pulse, respiration and O2 saturation values together with fear and pain scales after the application of virtual reality goggles 15 minutes before IT chemotherapy, and in the third measurement, electrodermal activity, pulse, respiration and O2 saturation values together with fear and pain scales will be evaluated within 30-60 minutes after IT chemotherapy treatment (when the sedation effect is over).
  Interventions: Other: Educational movie
- The group that received routine clinical care without any intervention (No Intervention): Measurements will be performed in three stages parallel to the treatment groups. In the first measurement; electrodermal activity, pulse, respiration and O2 saturation values together with fear and pain scales 30 minutes before IT chemotherapy treatment without any intervention, in the second measurement; In the second measurement, electrodermal activity, pulse, respiration and O2 saturation values together with fear and pain scales 15 minutes before IT chemotherapy, and in the third measurement, electrodermal activity, pulse, respiration and O2 saturation values together with fear and pain scales will be evaluated within 30-60 minutes after IT chemotherapy treatment (when the sedation effect is over).

INTERVENTIONS:
Other: Educational movie — There are three groups in this research. The 1st group will be shown an educational movie about intrathecal chemotherapy treatment before intrathecal chemotherapy treatment, the 2nd group will be shown a cartoon movie before intrathecal chemotherapy treatment, and the 3rd group will not receive any intervention before intrathecal chemotherapy treatment. In all groups, measurements will be made in parallel; fear and pain scales as well as electrodermal activity, pulse, respiration and O2 saturation values 30 minutes before IT chemotherapy treatment, in the second measurement; In the second measurement, electrodermal activity, pulse, respiration and O2 saturation values along with fear and pain scales 15 minutes before IT chemotherapy, and in the third measurement, electrodermal activity, pulse, respiration and O2 saturation values along with fear and pain scales will be evaluated within 30-60 minutes after IT chemotherapy treatment (when the sedation effect is over).
  Other Names: Cartoons; Without any intervention
  Arms: Group shown educational movie with virtual reality glasses; Group watching cartoons with virtual reality glasses

SUMMARY:
In this study, which is planned to be conducted in a randomized controlled experimental design, nonpharmacological methods (educational film shown with virtual reality goggles and cartoon shown with virtual reality goggles) applied to children aged 5-10 years who will receive intrathecal chemotherapy treatment before intrathecal chemotherapy treatment were evaluated. It is aimed to determine the effect on pre-procedure fear and post-procedure pain.

The study is planned to be conducted between November 2024 and November 2025. The population of the study will consist of children between the ages of 5-10 years who receive inpatient treatment in the Pediatric Hematology Clinic of Izmir Ege University Hospital (Health Practice and Research Center). Random sampling method and stratified randomization method will be used for sample selection. In the calculation of the sample size of the study, using G-Power 3.1.9.7 program; type 1 error (α) 0.05, power (1- β) 99% and Cohen's effect size (δ) 0.5, the sample size to represent the main mass was determined as 90 children for this study. However, when the dropout rate is set as 10% for data loss that may occur in the study, the minimum number to be reached for the study is targeted as 99 (intervention group 1 n=33, intervention group 2 n=33, control group n=33).

Research data will be collected after project acceptance. In all three groups, children and their parents will be informed before the study and their written and verbal consent will be obtained. Data will be collected by using the "Introductory Information Form", "Intervention Follow-up Form" and "Child Fear Scale (CFS)", "Wong Baker FACES (WB-FACES) Pain Rating Scale" and "Visual Analog Scale (VAS)" prepared by the researchers with the feedback of nurses, parents and children.

Statistical analyses will be performed using IBM SPSS Statistics 26.0 (IBM SPSS Statistics for Windows) package program. The significance level will be set as 0.05 in all analyzes. In the study, numerical data will be calculated using mean, standard deviation, median, minimum, maximum values and categorical data will be calculated using frequency and ratio values.

With the nonparametric Brunner-Langer model, the before-after change (group effect, before-after effect and interaction effect) of fear scores in the educational film, cartoon and control groups will be examined using R 3.3.1 software (R software, version 3.3.1, package: nparLD, R Foundation for Statistical Computing, Vienna, Austria; http://r-project.org). In order to visually examine this change, the 'relative effects' graph (since the nonparametric method is used) will be utilized.

When the Brunner-Langer model shows that the before-after change in the groups is not similar (interaction < 0.05), the before-after comparison in each group will be made separately with the Wilcoxon sign test, and the differences between the groups will be compared with the Kruskal-Wallis test by taking the after-before difference. After Kruskal-Wallis, pairwise comparisons will be made with the Dunn test, and then Bonferroni correction will be used for p values. The agreement between the measurements of Nurses, Parents and Children will be evaluated by Intraclass Correlation (ICC) analysis.

ELIGIBILITY:
Inclusion Criteria:

* 5-10 years old
* Family's acceptance to participate in the research
* The child's willingness to participate in the research
* Absence of a pancytopenic period
* No sensory loss
* Developed language skills/no communication problems
* Lack of a psychological diagnosis Cognitive abilities are developed in an age-appropriate manner
* Having not used any anelgesic drug in the last four hours

Exclusion Criteria:

* The child has an infection that requires isolation
* The child wears glasses
* Child removes virtual reality goggles applied before intrathecal chemotherapy treatment
* The child does not want to fill in the scales after the application
* The child or parent wants to leave the study
* The child has a physical and psychological deficit that prevents him/her from wearing the glasses that will be worn on his/her head in order to watch virtual reality

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Pain | Measurements will be performed 30 minutes before intrathecal chemotherapy (without any intervention to the child), 15 minutes before intrathecal chemotherapy (after application of virtual reality goggles), and 30-60 minutes after IT chemotherapy (after t
  Wong Baker FACES (WB-FACES) Pain Rating Scale: The WB-FACES scale was first developed by Donna Wong and Connie Baker in 1981 and updated in 1983. This scale is used for pain assessment in children between the ages of 3 and 18. A simple tool including five different facial expressions was created by taking into account the way children express their pain. This scale is used to determine the level of pain in children aged 3-18 years. It contains a total of 6 facial expressions and provides a rating scale between 0-10. It does not require word or numeric values and is reported to be a reliable and valid measurement tool in the evaluation of acute pain. As the score obtained from the scale increases, the severity of pain increases and as the score decreases, the severity decreases.
Pain | Measurements will be performed 30 minutes before intrathecal chemotherapy (without any intervention to the child), 15 minutes before intrathecal chemotherapy (after application of virtual reality goggles), and 30-60 minutes after IT chemotherapy (after t
  Visual Analog Scale (VAS): The Visual Analog Scale (VAS), developed by Price et al. (1983), is one of the widely used tools for pain assessment in children. The VAS is characterized by its ease of use and simple structure. It allows children to mark their pain on a line or a line. The scale consists of a line at one end indicating no pain and a line at the other end indicating excruciating pain. By marking their own pain, children determine how much pain they feel.
Fear | Measurements will be performed 30 minutes before intrathecal chemotherapy (without any intervention to the child), 15 minutes before intrathecal chemotherapy (after application of virtual reality goggles), and 30-60 minutes after IT chemotherapy (after t
  Child Fear Scale: The Facial Expressions of Fear Scale was developed by McKinley et al. (2003) as "The Faces Anxiety Scale" to measure the fear or anxiety of adults hospitalized in the intensive care unit. The Child Fear Scale was developed by McMurty et al. (2011) by adapting the Facial Expressions of Fear Scale to children. The scale consists of five drawn facial expressions ranging from a neutral expression (0=no anxiety) to a frightened face (4=severe anxiety) and can be easily evaluated by researchers and health professionals who provide care/intervention to children. The scale was translated into Turkish by Gerçeker et al. in 2018. Content validity is the most frequently used method in the validity of measurement tools. The content validity index of the CQS was found to be 0.89.

SECONDARY OUTCOMES:
Electrodermal activity | Measurements will be performed 30 minutes before intrathecal chemotherapy (without any intervention to the child), 15 minutes before intrathecal chemotherapy (after application of virtual reality goggles), and 30-60 minutes after IT chemotherapy (after t
  Electrodermal activity device: An electrodermal activity device is a biometric measurement tool that measures changes in electrical conductivity on the skin surface. This device is often used to study a person's emotional and physiological responses. In particular, EDA reflects changes in the skin's conductivity due to the activity of sweat glands, which is associated with states such as stress, fear, excitement or arousal. In this study, the electrodermal activity device will be used simultaneously with the Child Fear Scale to measure the fear experienced by children before, during and after intrathecal chemotherapy treatment.
Pulse | Measurements will be performed 30 minutes before intrathecal chemotherapy (without any intervention to the child), 15 minutes before intrathecal chemotherapy (after application of virtual reality goggles), and 30-60 minutes after IT chemotherapy (after t
  Pulseoximeter Calibrated pulseoximeter device will be used for pulse and O2 saturation measurements of children.
Respiration | Measurements will be performed 30 minutes before intrathecal chemotherapy (without any intervention to the child), 15 minutes before intrathecal chemotherapy (after application of virtual reality goggles), and 30-60 minutes after IT chemotherapy (after t
  Pulseoximeter Calibrated pulseoximeter device will be used for pulse and O2 saturation measurements of children.
O2 saturation | Measurements will be performed 30 minutes before intrathecal chemotherapy (without any intervention to the child), 15 minutes before intrathecal chemotherapy (after application of virtual reality goggles), and 30-60 minutes after IT chemotherapy (after t
  Pulseoximeter Calibrated pulseoximeter device will be used for pulse and O2 saturation measurements of children.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, BORNOVA, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No